CLINICAL TRIAL: NCT02270892
Title: Evaluation of the Ulthera® System for Lifting of the Buttock
Brief Title: Ultherapy for Buttock Lift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-142
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2017-05

CONDITIONS: Buttock Ptosis
Keywords: Ulthera, Ulthera System, Ultherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Left side Ulthera treatment
  Interventions: Device: Ulthera treatment
- Group B (Active Comparator): Right side Ulthera treatment
  Interventions: Device: Ulthera treatment

INTERVENTIONS:
Device: Ulthera treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy, Ulthera System Treatment

SUMMARY:
Up to 24 subjects will be enrolled and treated. Enrolled subjects will receive two Ulthera® treatments, 90 days apart. Follow-up visits will occur at 90, 180, and 270 days following the last treatment. Study images will be obtained pre-treatment, immediately post-treatment, and at each follow-up visit.

DETAILED DESCRIPTION:
This study is a prospective, single-blinded, randomized, split-body clinical study to be conducted at one clinical site. Investigator will assess baseline buttock ptosis to confirm subject eligibility.

Enrolled subjects meeting all entrance criteria and who are confirmed to be eligible for study treatment will be randomized/assigned into one of two treatment groups: "Right side treated" and "Left side treated". All subjects will receive two, single-sided, dual-depth Ultherapy® treatments using the 4-4.5mm and 7-3.0mm transducers at 0.90J and 0.30J, respectively. Standardized images will be taken using standard 2D and Vectra 3D digital imaging systems. Subjects completing all study visits will be given the option of receiving two balancing treatments, 90 days apart, and will be required to complete one study visit at 90 days following the last balancing treatment. Quantititative and qualititative assessment of pre- versus post-treatment buttock ptosis will be completed for each post-treatment time point. Subjects will also complete a questionnaire at each study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age 18 to 65 years.
2. Subject in good health.
3. Mild to moderate buttock ptosis based on Investigator evaluation.
4. BMI <25.
5. No history of weight gain or loss of greater than 10 pounds within the past year.
6. No planned weight loss or gain for the duration of the study.
7. No pregnancy within the past year.
8. Willingness to refrain from use of aspirin, Ibuprofen, Naproxen or any other NSAID prior to each study treatment and chronic use during the entire post-treatment study period. If a chronic user, a washout period of 4 weeks is required prior to study treatment #1. Washout period for limited acute NSAID use, i.e., a maximum of 2-3 doses, is required in the 2 weeks prior to any study treatment visit.
9. No immunosuppressive therapy, e.g., oral steroid treatment, within the past 4 weeks and during the entire post-treatment study period. Washout period, if recent use, for 4 weeks prior to study treatment #1.
10. Subject must desire improvement of her buttock ptosis as demonstrated by a Dissatisfaction response on a baseline Patient Satisfaction Questionnaire, i.e., Dissatisfied, Neither Satisfied or Dissatisfied, Slightly Satisfied, Satisfied, Very Satisfied.
11. Willingness to refrain from receiving spray tans or using self-tanning lotions from mid-thigh to waist within 2 weeks of any study assessments for the duration of the trial.
12. Willingness to avoid as much as possible, direct and prolonged sun exposure from mid-thigh to waist for the duration of the study.
13. Willingness to refrain from topical steroid use, tretinoin, caffeine cream and other prescription or over-the-counter cellulite reduction topicals to the affected area 2 weeks prior to study treatment #1 and for the duration of the study period.
14. Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
15. Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
16. Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Baseline Visit and be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

    1. Postmenopausal for at least 12 months prior to study;
    2. Without a uterus and/or both ovaries; or
    3. Bilateral tubal ligation at least six months prior to study enrollment.
17. Absence of physical or psychological conditions unacceptable to the investigator.
18. Willingness and ability to provide written consent for study-required photography and adherence to photography procedures.
19. Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

1. Radiofrequency, CoolSculpting, liposuction, other energy-based treatment in the area to be treated for body contouring, fat reduction, improvement of cellulite, or reduction of buttock ptosis within 1 year prior to study participation or during the study.
2. Short-wave or massage therapy in the area to be treated for treatment of cellulite or buttock ptosis within 3 months prior to study participation or during the study.
3. BMI greater than or equal to 25.
4. Presence of an active systemic or local skin disease that may affect wound healing.
5. Excessive subcutaneous fat in the area to be treated.
6. Excessive skin laxity on the area to be treated.
7. Severe buttock ptosis.
8. Significant scarring or tattoos in the area to be treated that would interfere with assessing results.
9. Open wounds or lesions in the area to be treated.
10. Inability to understand the protocol or to give informed consent.
11. History of chronic drug or alcohol abuse.
12. History of autoimmune disease.
13. Has a known allergy or a known contraindication to ketorolac tromethamine (Toradol).
14. Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
15. Subjects who anticipate the need for inpatient surgery or overnight hospitalization during the study.
16. Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
17. Concurrent enrollment in any study involving the use of investigational devices or drugs.
18. Current smoker or history of smoking in the last 5 years.
19. Current user of any nicotine-containing products, e.g., e-cigarettes, Nicorette gum, nicotine patches, etc.
20. History of the following cosmetic treatments in the area to be treated:

    1. Skin tightening procedure within the past year;
    2. Buttock implants;
    3. Buttock fillers (e.g., silicone, semi-permanent or permanent fillers or autologous fat injections);
    4. Fat emulsifiers;
    5. Injections for the treatment of cellulite.
21. History of using the following prescription medications:

    1. Accutane or other systemic retinoids within the past 6 months;
    2. Topical retinoids, tretinoin, caffeine cream and other prescription or over-the-counter cellulite reduction topicals within the past 2 weeks;
    3. Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix);
    4. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2016-07-22 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
90-day quantitative buttock lift | 90 days following last treatment
  Post-treatment change from baseline in protocol-defined buttock measurements:
  * ϒ (gamma) angle: The angle between the turning point between the gluteal sulcus line and the thigh;
  * β (beta) angle: The angle from the midpoint of the lateral thigh along the gluteal-sulcus line and the most posterior point of the buttock.
180-day quantitative buttock lift | 180 days following last treatment
  Post-treatment change from baseline in protocol-defined buttock measurements:
  * ϒ (gamma) angle: The angle between the turning point between the gluteal sulcus line and the thigh;
  * β (beta) angle: The angle from the midpoint of the lateral thigh along the gluteal-sulcus line and the most posterior point of the buttock.
270-day quantitative buttock lift | 270 days following last treatment
  Post-treatment change from baseline in protocol-defined buttock measurements:
  * ϒ (gamma) angle: The angle between the turning point between the gluteal sulcus line and the thigh;
  * β (beta) angle: The angle from the midpoint of the lateral thigh along the gluteal-sulcus line and the most posterior point of the buttock.

SECONDARY OUTCOMES:
90-day qualitative improvement in buttock ptosis | 90 days following last treatment
  Determined by a masked, qualitative assessment of 2D photographs compared to baseline.
180-day qualitative improvement in buttock ptosis | 180 days following last treatment
  Determined by a masked, qualitative assessment of 2D photographs compared to baseline.
270-day qualitative improvement in buttock ptosis | 270 days following last treatment
  Determined by a masked, qualitative assessment of 2D photographs compared to baseline.
90-day Clinician Buttock Improvement Scale (CBIS) | 90 days following last treatment
  CBIS assessing overall aesthetic improvement based on a 5-point scale, rating improvement from the pre-treatment appearance:
  * 1=very much improved
  * 2=much improved
  * 3=improved
  * 4=no change
  * 5=worse
180-day Clinician Buttock Improvement Scale (CBIS) | 180 days following last treatment
  CBIS assessing overall aesthetic improvement based on a 5-point scale, rating improvement from the pre-treatment appearance:
  * 1=very much improved
  * 2=much improved
  * 3=improved
  * 4=no change
  * 5=worse
270-day Clinician Buttock Improvement Scale (CBIS) | 270 days following last treatment
  CBIS assessing overall aesthetic improvement based on a 5-point scale, rating improvement from the pre-treatment appearance:
  * 1=very much improved
  * 2=much improved
  * 3=improved
  * 4=no change
  * 5=worse
90-day Subject Buttock Improvement Scale (SBIS) | 90 days following last treatment
  SBIS assessing overall aesthetic improvement based on a 5-point scale, rating improvement from the pre-treatment appearance:
  * 1=very much improved
  * 2=much improved
  * 3=improved
  * 4=no change
  * 5=worse
180-day Subject Buttock Improvement Scale (SBIS) | 180 days following last treatment
  SBIS assessing overall aesthetic improvement based on a 5-point scale, rating improvement from the pre-treatment appearance:
  * 1=very much improved
  * 2=much improved
  * 3=improved
  * 4=no change
  * 5=worse
270-day Subject Buttock Improvement Scale (SBIS) | 270 days following last treatment
  SBIS assessing overall aesthetic improvement based on a 5-point scale, rating improvement from the pre-treatment appearance:
  * 1=very much improved
  * 2=much improved
  * 3=improved
  * 4=no change
  * 5=worse
90-day Patient Satisfaction Questionnaire (PSQ) | 90 days following last treatment
  Patient satisfaction with treatment assessed based on completion of a PSQ.
180-day Patient Satisfaction Questionnaire (PSQ) | 180 days following last treatment
  Patient satisfaction with treatment assessed based on completion of a PSQ.
270-day Patient Satisfaction Questionnaire (PSQ) | 270 days following last treatment
  Patient satisfaction with treatment assessed based on completion of a PSQ.
Balancing treatment 90-day Patient Satisfaction Questionnaire (PSQ) | 90 days following last balancing treatment
  Patient satisfaction with treatment assessed based on completion of a PSQ.
Balancing treatment 90-day Subject Buttock Improvement Scale (SBIS) | 90 days following last balancing treatment
  SBIS assessing overall aesthetic improvement based on a 5-point scale, rating improvement from the pre-treatment appearance:
  * 1=very much improved
  * 2=much improved
  * 3=improved
  * 4=no change
  * 5=worse
Balancing treatment 90-day Clinician Buttock Improvement Scale (CBIS) | 90 days following last balancing treatment
  CBIS assessing overall aesthetic improvement based on a 5-point scale, rating improvement from the pre-treatment appearance:
  * 1=very much improved
  * 2=much improved
  * 3=improved
  * 4=no change
  * 5=worse
Balancing treatment 90-day quantitative buttock lift | 90 days following last balancing treatment
  Post-treatment change from baseline in protocol-defined buttock measurements:
  * ϒ (gamma) angle: The angle between the turning point between the gluteal sulcus line and the thigh;
  * β (beta) angle: The angle from the midpoint of the lateral thigh along the gluteal-sulcus line and the most posterior point of the buttock.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Misell, PhD, Study Director — Ulthera, Inc
Locations (1):
- Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc., La Jolla, California, United States